CLINICAL TRIAL: NCT02934672
Title: KineSpring® System Patient Preference Study
Status: Completed | Type: Observational
Sponsor: Moximed (Industry)
Responsible Party: Sponsor
Other Study IDs: 102392
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Survey — Internet panelists, who self-reported that they or another adult in their household has osteoarthritis, were sent an email invitation to the survey site.

SUMMARY:
The primary objectives of the survey are to obtain patient preference information that can be useful during the benefit-risk assessment of the KineSpring System.

DETAILED DESCRIPTION:
Well-established, quantitative research methods were employed to understand the relative importance of effectiveness, safety, and other characteristics of orthopedic surgical treatments and develop a benefit-risk model to inform regulatory decision making.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 25 - 80 years
* Diagnosed with osteoarthritis in the knee
* Experience pain in the knee of greater than or equal to a "4" on a "0 - 10" scale, where 0 means not at all painful and 10 means extremely painful
* Experience knee pain at least once a week
* Previously failed non-surgical treatments for knee OA pain
* Pass a security screen

Exclusion Criteria:

* Do not suffer or has not been diagnosed with knee osteoarthritis
* Has had knee surgical intervention involving an implant or a prosthesis (i.e. total knee replacement, unicompartmental knee arthroplasty, high tibial osteotomy)

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females aged 25 to 80 years old diagnosed with osteoarthritis in the knee
Sampling Method: Non-Probability Sample
Enrollment: 323 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Patient preferences for knee osteoarthritis surgical procedures | At time of survey
  Patient preference for knee osteoarthritis surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Yamut, Study Director — Moximed

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moorman CT 3rd, Kirwan T, Share J, Vannabouathong C. Patient Preferences Regarding Surgical Interventions for Knee Osteoarthritis. Clin Med Insights Arthritis Musculoskelet Disord. 2017 Sep 20;10:1179544117732039. doi: 10.1177/1179544117732039. eCollection 2017. PMID 28974919